CLINICAL TRIAL: NCT05791500
Title: Investigation of Undergraduate Lifestyle Such as Diet and Exercise and Its Interventions on Relevant Factors on Campus
Brief Title: Investigation of Undergraduate Lifestyle and Its Related Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Junjie Wu, Principal Investigator, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20221011-3
Record Dates: First submitted 2023-02-28; First posted 2023-03-30 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Life Style, Healthy; Diet, Healthy; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- lifestyle intervention group (Experimental): People in intervention group are required to have a daily work and rest time of 7-8 hours, adjusted according to their original work and rest, but no later than 9:00 to get up and 23:00 to fall asleep; change their intimate clothes every day and clean themselves at least twice a day（mainly including brushing their teeth and washing their faces at least twice in the morning and evening, and showering once）The bed is guaranteed to sun/wash the quilt once a month, the sheets are changed twice a week in spring and autumn, and once a month in winter. The desk in the dorm is arranged neatly and orderly, the study and daily necessities are sorted and placed, at least there is place for office and study, the bed is clean and tidy, no garbage, no dirt. It is required to upload the hygiene situation of the bedroom (including the desk and the bed) once a week, and take a photo every time the bedding is changed.
  Interventions: Behavioral: lifestyle intervention
- lifestyle control group (No Intervention): This group doesn't conclude any intervention measures.But the data of participants is obtained at the same time as the intervention group.
- dietary habits intervention group (Experimental): Before the interventions,data such as dietary health scores which includes Dietary Quality Index(DQI) ,score based on dietary health questionaire and so on are collected.Then people in the intervention group are gathered to participate in dietary health education lectures,after which the data such as DQI will be obtained again.
  Interventions: Behavioral: lifestyle intervention
- dietary habits control group (No Intervention): This group doesn't conclude any intervention measures.But the data of participants is obtained at the same time as the intervention group.
- physical activity intervention Group A-jogging (Experimental): People in the Group A-jogging need to training at least 4 times a week, each time at least 50 minutes for boys and at least 40 minutes for girls, for 4 months. Before the experiment, students in the Group A-jogging learned the basic movements and complete sets of movements of this exercise prescriptions.
  Interventions: Behavioral: lifestyle intervention
- physical activity intervention Group B-rope skipping (Experimental): People in the Group B-rope skipping need to training at least 4 times a week, each time at least 50 minutes for boys and at least 40 minutes for girls, for 4 months. Before the experiment, people in the Group B-rope skipping learned the basic movements and complete sets of movements of this exercise prescriptions.
  Interventions: Behavioral: lifestyle intervention
- physical activity Control Group (No Intervention): This group doesn't conclude any intervention measures.But the data of participants is obtained at the same time as the intervention group.

INTERVENTIONS:
Behavioral: lifestyle intervention — dietary behavior interventions:through a couple of dietary health education lectures physical activity interventions:through at least an offline teaching and jump rope or jog regularly and quantitatively life schedule and habits intervention group: live in a regular and healthy life habit and last at least 4 months
  Arms: dietary habits intervention group; lifestyle intervention group; physical activity intervention Group A-jogging; physical activity intervention Group B-rope skipping

SUMMARY:
It is already known that lifestyle is closely related to human health, disease formation, learning and work efficiency. Although there have been relevant researches on lifestyle, there is no research on the current situation of college students' lifestyle and its correlation with their studies; In addition, how to effectively and scientifically intervene unhealthy lifestyles and observe the sustainability of the intervention effect has not been reported. Therefore, this research takes the students in Zhejiang University of Traditional Chinese Medicine as the research object to carry out a survey, understand the current situation of their lifestyle, analyze the influence of gender, major, grade and education on their lifestyle, and explore the correlation between lifestyle and academic performance; And then the targeted intervention is to be carried out against the unhealthy lifestyle factors in order to observe the intervention effect and its sustainability

DETAILED DESCRIPTION:
1、Population：Domestic undergraduates, no major diseases, lower grades (freshman, sophomore, junior, senior), are not receiving any special treatment or in a state of intervention.

2、intervention：

1. Dietary habits intervention group:

   (1)．Canteen intervention
   1. Select some shops from the dining hall of Zhejiang Chinese Medical University, and randomly set them into the control group and the intervention group by drawing lots. Before the intervention, take photos of all kinds of food in the shop and collect their monthly sales data, calculate their caloric value according to the Chinese food composition database, score each dish through DQI-I(Dietary Quality Index-International), and make food labels.
   2. Put up food labels on the menu of the intervention group's door shop, and do not paste food labels on the control group's door shop. A one month intervention experiment will be carried out after ensuring that there won't be any other activities like discount or any changes to the dishes sold in the shop during the experiment.
   3. After the intervention, the sales data of various kinds of food products in the shops of the control group and the intervention group in November were counted again.

   (2)． Crowd intervention 4、80 volunteers (α =0.05、1- β =0.9, SD(standard deviation)= 6.79, δ =5),are recruited in Zhejiang Chinese Medical University by posting posters in the dining hall and in the form of posters spread by QQ or WeChat(two popular social media platforms) , and divide them into the control group and the intervention group by randomly drawing lots, Before the intervention, the baseline dietary health data of volunteers are collected by food pictures taken within three days and filling in the KABP(Knowledge,Attitude,Belief,Practice) questionnaire for college students' health literacy: food pictures are scored according to the International Dietary Quality Index (DQI-I), and then the dietary health literacy data of college students (including dietary health level, dietary health knowledge and dietary health attitude) is obtained through the Knowledge-Attitude,Belief-Practice(KABP) model based questionnaire for dietary health.

   5、lay down dietary health education measures based on KABP model, which emphasizes on improving people's belief in diet health (In the course, students can be taught the dangers of unhealthy diet through some videos, and it is not difficult to form a healthy diet, and students can realize the benefits of healthy diet, so that students can understand the importance of healthy diet, which will improve their attitude and brief towards dietary health.), The course topics may include reasonable diet to lose weight, how to carry out the nutrition matching of three meals, and the classification of unhealthy food. And the courses are scheduled on every Wednesday afternoon for four times.

   6、After the four courses, the students were asked to upload the pictures of the food they had eaten for three days again, fill in the KAP(Knowledge,Attitude,Practice) questionnaire on dietary health again, and we will calculate the total score and analyse the differences
2. Exercise habit intervention group:

   1．Intervention object： A total of 90 healthy student volunteers (mainly sophomores and juniors) are recruited from Zhejiang University of Traditional Chinese Medicine.There are 30 people in the blank control group and 60 people in the intervention group (30 people in the running group and 30 people in the jumping rope group).Numbers will be adjusted depending on recruitment.

   2. Theory teaching The PE teacher is invited to give a theoretical teaching before the sports training intervention to explain the benefits, functions and methods of physical exercise.

   3. Athletic training The volunteers are randomly assigned to three groups (blank control group, running group and rope skipping group). The two groups of intervention students are given running exercise and rope skipping exercise training at least 4 times a week, each time at least 50 minutes for boys and at least 40 minutes for girls, for a consecutive semester. Before the experiment, students in the two intervention groups learn the basic movements and complete sets of movements of the two exercise prescriptions , so as to ensure the training quality in the experiment period and reduce injuries.

   Remarks: The training intensity of the exercise intervention will be strengthened according to the actual situation in the middle and later period of the intervention; Exercise interventions are expected to use applications and other forms of objective data collection and monitoring.

   4．index testing： Students are tested uniformly before the intervention, Selection of college students' body mass index (BMI,kg/m^2), the main life/physiological indexes (blood pressure, heart rate, breathing, etc.) in succession, crook proneness, standing long jump, pull-ups (male)/sit-ups (female) and 1000 - meter run (male) / 800 - meter run (female), 50 meters, body fat index to assess students' flexibility quality, power quality, endurance quality. At the end of the experiment, students are tested again. Finally, the scores of each physical test are analyzed and compared between the intervention group and the blank control group, and the scores of the last physical test before and after the intervention are analyzed and compared between the two groups.
3. Life Schedule And Habits Intervention Group:

   1. Recruit experimental volunteers（The specific method is to send advertisements online,place recruitment roll-ups at the entrance of the canteen, and release promotional posters in the WeChat and grade groups），and randomly divide them into three groups: Life Schedule Intervention Group, Lifestyle Intervention Group and Control Group.Before the intervention experiment, all volunteers are required to fill out a questionnaire to collect the current status and relationship between the lifestyle and academic performance of the volunteers before the intervention experiment.
   2. Life Schedule and habits Intervention Group requires the volunteers to have a daily work and rest time of 7-8 hours, adjusted according to their original work and rest, but no later than 9:00 to get up and 23:00 to fall asleep; Volunteers are asked to record daily schedule and approximate time of falling asleep and getting up. Upload the screenshots of their mobile phones and schedules every week. In the same time, volunteers are required to change their intimate clothes every day and clean themselves at least twice a day（mainly including brushing their teeth and washing their faces at least twice in the morning and evening, and showering once）The bed is guaranteed to sun/wash the quilt once a month, the sheets are changed twice a week in spring and autumn, and once a month in winter. The desk in the dorm is arranged neatly and orderly, the study and daily necessities are sorted and placed, at least there is place for office and study, the bed is clean and tidy, no garbage, no dirt. It is required to upload the hygiene situation of the bedroom (including the desk and the bed) once a week, and take a photo every time the bedding is changed.
   3. Before and during the intervention, the researchers shared relevant popular science videos, public accounts, articles, etc. on factors such as lifestyle and life schedule to the Life Schedule Intervention Group, Lifestyle Intervention Group. The intervention lasts one semester. The control group did not do the above intervention treatment, but still carried out relevant data collection.

After the end of the intervention experiment, all volunteers (including the intervention group and the control group) filled in the questionnaire to collect the current situation and relationship between the volunteers' lifestyle and academic performance before the intervention experiment. Two months after the end of the intervention, the current lifestyle status of all volunteers is re-collected, and the effect of the intervention is assessed on the current status and relationship between the intervention and lifestyle, academic performance, and each other.

3、Comparison：No interventions above, only the questionnaire is required to collect basic information.

4、Outcome：The level of health status of college students (diet, exercise, psychology, work and rest, bad habits), academic level 5、Study design：randomised controlled trials

ELIGIBILITY:
Inclusion Criteria:

- Undergraduates, lower grades (freshman, sophomore, junior, senior)

Exclusion Criteria:

- major illnesses, are receiving some special treatment or are themselves in a state of intervention

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
GPA(Grade Point Average) | four months
  participators' academic performance
lifestyle index | four months
  index of participators' living habits
Physical body gat and key vital/physiological index such as weight(kilogram),height(meter) | four months
  index of participators' physical quality
University students' physical exercise consciousness, habit, type and its influencing factors questionnaire | four months
  performance of participators' physical activity and its related factors
University students' dietary health score | four months
  collect three days' of food pictures and quantize them to get a dietary health score
University students' dietary behavior | four months
  through a dietary health KABP(Knowledge,Attitude,Belief,Practice) questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Qinghua Sun, professor, Study Director — Zhejiang Chinese Medical University School of Public Health
Locations (1):
- Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China